CLINICAL TRIAL: NCT02787278
Title: A Prospective, Randomized, Double-blinded Phase IIa Clinical Trial to Investigate the Safety and Efficacy of Two Doses of SP-8203 in Patients With Ischemic Stroke Requiring rtPA Standard of Care
Brief Title: Safety and Efficacy of Two Doses of SP-8203 in Patients With Ischemic Stroke Requiring rtPA
Acronym: SP-8203-2001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-8203-2001
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Ischemic Stroke
Keywords: rtPA; Intracranial hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages | interventions — otaplimastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SP-8203 High dose group (Experimental): SP-8203 160mg (80mg/dose twice a day for three days)
  Interventions: Drug: SP-8203 High dose
- SP-8203 Low dose group (Experimental): SP-8203 80mg (40mg/dose twice a day for three days)
  Interventions: Drug: SP-8203 Low dose
- Placebo group (Placebo Comparator): Placebo group: twice a day for three days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-8203 High dose — High-dose group: 160mg will be intravenously administered as 80mg/dose twice daily (intervals of 12 hours).
  Other Names: SP-8203 is produced by Shin Poong Pharmaceutical company
  Arms: SP-8203 High dose group
Drug: SP-8203 Low dose — Low dose group: 80mg will be intravenously administered as 40mg/dose twice daily (intervals of 12 hours).
  Other Names: SP-8203 is produced by Shin Poong Pharmaceutical company
  Arms: SP-8203 Low dose group
Drug: Placebo — Same dosage of SP8203. Placebo will be intravenously administered twice daily (intervals of 12 hours)
  Arms: Placebo group

SUMMARY:
The current study aims to evaluate the safety of SP-8203, designing in two stages (stage-1, stage-2) to evaluate the safety and efficacy of the combination therapy of SP-8203 and rtPA for the occurrence of cerebral hemorrhage in patients with acute ischemic stroke receiving rtPA standard of care.

DETAILED DESCRIPTION:
As the standard procedure of rtPA therapy, rtPA will be injected intravenously using a device like infusion pump. When reperfusion is not achieved in spite of rtPA therapy, endovascular therapy can be performed according to the judgment of a site investigator.

Stage 1-The trial will be conducted with 11 subjects participating in an open label design manner. Subjects with neurologic deficit of ≥4 point and ≤10 points on NIHSS score will be given SP-8203, 80mg/dose, a total of 6 times at intervals of 12 hours. For the first administration of SP-8203, it should be administered within 30 minutes from the initiation of rtPA administration via a vein route different from one via which rtPA is injected.

Thereafter, the subject will be transferred to MRI scanning room to have brain MRI and MRA performed, and brain CT will be performed to check the occurrence of intracranial hemorrhage at 24 hours after complete administration of the first dose of SP-8203. The subject will be closely monitored by research staff daily from the day of first administration of SP-8203 (Day 0) to Day 5. Brain MRI and MRA will be followed up after the last administration of SP-8203 on Day 5. The subject will make a visit on Day 14 to have his/her neurologic symptoms checked, after which subject's participation in the trial will be completed.

*The DSMB (Date Safety Monitoring Board) meeting will be held, to decide whether to proceed with Stage 2 or not, based on the results of Stage 1.

Stage 2- A total of 69 subjects will be enrolled in double-blind, randomized and parallel design with 23 subjects assigned to low-dose (40mg/dose, 80mg/ day) SP-8203 group, high-dose (80mg/dose, 160mg/day) SP-8203 group or placebo group, respectively.

If a subject, who is able to be enrolled in Stage 2, has neurological deficit of ≥4 point on NIHSS score and give patient's consent to participate in the trial, randomization will be performed and each treatment arm (one of three) will be assigned. The subject will receive the Investigational products a total of 6 times, with 12 hours intervals. Blood sample will be taken after the sixth administration of the Investigational product for pharmacokinetic and pharmacodynamics analysis. For pharmacokinetic analysis , blood sample will be taken at 0, 30, and 120 minutes after the complete sixth administration of the investigational products. For pharmacodynamics analysis, blood sample will be taken at between 24 to 48 hours after the first administration, at 0 minute after the sixth administration and at 4th week visit.

As with Stage 1, the subject will have brain MRI and MRA performed after the administration of investigational product, and brain CT will be performed at 24 hours after completion of the first administration of investigational products.

Brain MRI and MRA will be followed-up on Day 5, similarly to Stage 1. However, in Stage 2, the subject will make a visit for close monitoring for patient's neurological condition at 4th week and 12th week. Thereafter, all the procedures of the clinical trial will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1-specific Criteria Patients with neurologic deficit of ≥4 points and ≤10 points by NIHSS score.

Stage 2-specific Criteria Patients with neurologic deficit of ≥4 points by NIHSS score.

Common Criteria for Stage 1 and Stage 2

1. Adults aged ≥19 years and ≤80 years.
2. Subjects fulfilling the criteria for rtPA therapy. ① Subjects who can receive rtPA therapy within 4.5 hours after the onset of early symptoms of acute ischemic stroke.

   ② Subjects requiring rtPA therapy according to the judgment of a neurologist.
3. Subjects available for brain MRI (DWI, GRE/SWI [Susceptibility Weighted Imaging], FLAIR, MRA) scanning
4. Subjects who consent to participate in this trial.

Exclusion Criteria:

1. Patients with systemic allergic diseases or hypersensitivity to specific drugs.
2. Patients have condition as follows:

<!-- -->

1. Patients who were diagnosed with acute myocardial infarction (AMI) within the last 6 months.
2. Patients who had arrhythmia causing symptoms such as dyspnea or palpitation within the last 6 months.
3. Patients showing the following abnormal ECG findings in stable condition at screening:

   * The range of pulse rate - below 60/min or above 120/min

     * 2nd or 3rd degree AV(Atrioventricular) block indicated in ECG

       * Congenital or acquired QT syndrome indicated in ECG

         ④ Pre-excitation syndrome indicated in ECG

         3) Patients with severe heart failure of NYHA(New York Heart Association) Class III or Class IV.

NYHA classification of heart failure defined as:

Class I: patients with no limitation of activities; they suffer no symptoms from ordinary activities.

Class II: patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion.

Class III: patients with marked limitation of activity; they are comfortable only at rest.

Class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on.

4) Patients with fever (≥ 38℃) or infection signs which require antibiotics at screening 5) Patients with pulmonary diseases (asthma, COPD[Chronic Obstructive Pulmonary Disease ], and active tuberculosis etc.) who have being recently been treated more than 1 month at screening, 6) Patients showing the following hematological findings: Patients with decreased hemoglobin (Hb< 10g/dL), decreased platelet count (PLT< 100,000/mm3) or hematocrit of <25% in complete blood count .

7) Patients who have undergone hemodialysis and/or treatments due to nephropathies, acute or chronic renal failure at screening.

8) Patients with a cancer in following conditions: diagnosed within 6 months before the screening time, or any treatment for cancer within the previous 6 months, or with recurrent/ metastatic cancer 9) Pregnant and breast-feeding women. However, women of childbearing age can participate in the trial only when non-pregnancy is confirmed. Woman of childbearing age is defined as woman who is not definitely menopause and did not receive a surgical contraception 10) Patients who do not consent to use double barrier contraception during the trial period.

11) Patients who have participated in other clinical trials of other drugs within the past 3 months. However, if they participated in observational studies and did not take drugs, they can participate in this trial.

12) Patients who cannot participate in the trial according to the judgment of investigators.

13) Patients with contraindication for the use of rtPA as shown in the below. [Contraindication for the Use of rtPA] A. Patients with hypersensitivity to gentamycin

B. rtPA should not be administered when the risk of bleeding is high as follows:

i. Patients who suffered from significant hemorrhagic diseases within the past 6 months or with known hemorrhagic diathesis.

ii. Patients receiving oral anticoagulants such as warfarin sodium (INR>1.3). iii. Patients with apparent hemorrhage or recent serious or risky hemorrhage. iv. Patients with the past history of tumor, aneurysm, or central nervous system damage such as intracranial or intraspinal operation.

v. Patients with hemorrhagic retinopathy, diabetes accompanied with visual disturbance or other ophthalmic hemorrhage.

vi. Patients who underwent prolonged or traumatic cardiopulmonary resuscitation (>2 minutes), obstetrical delivery or recently incompressible vascular puncture within the recent 10 days.

vii. Patients with uncontrollable severe arterial hypertension. viii. Patients who have underwent major surgery for the recent 3 months or had recently significant trauma including all the trauma cases related with acute myocardial infarction or head trauma.

ix. Patients with bacterial endocarditis and pericarditis. x. Patients with acute pancreatitis. xi. Patients confirmed to have records of ulcerative gastrointestinal diseases, esophageal varix, aneurysm or arteriovenous malformation for the recent 3 months.

xii. Patients with severe liver diseases including hepatic failure, liver cirrhosis, portal hypertension (esophageal), or active hepatitis.

C. Patients with mild neurologic deficit of <4 points on the NIHSS, or severe condition of >25 points on the NIHSS.

D. Patients with seizure at onset of stroke. E. Patients with clinical presentation which suggests a subarachnoid hemorrhage, even if initial CT scan is normal.

F. Patients who received heparin and have elevated active partial thromboplastin time (aPTT) within 48 hours before the onset of stroke.

G. Patients who has history of stroke or had head injury within the recent 3 months.

H. Patients with systolic blood pressure of >185mmHg or diastolic BP of >110mmHg, or who require aggressive treatment (intravenous administration) to reduce BP to the limits.

I. Patients with blood glucose level of <50mg/dL or >400mg/dL.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06-05 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
The ratio of the incidence of parenchymal hematoma observed on brain CT | Brain CT should be performed at 24 ± 3 hours after the complete administration of the first dose of IP. (Screening, Baseline ,Day 0, Day 1)
  Incidence of parenchymal hematoma observed on brain CT performed at 24 hours in accordance with European Cooperative Acute Stroke Study (ECASS) I and II criteria

SECONDARY OUTCOMES:
Incidence rate of serious adverse events | Follow up period is 30 days after the last visit.
  Incidence rate of serious adverse events
Neurologic outcomes evaluated by modified Rankin Scale (mRS) | Screening, Baseline, Day 0, Day 5, Week 12, Early Termination
  Neurologic outcomes evaluated by modified Rankin Scale (mRS)
Incidence rate symptomatic intracranial hemorrhage (sICH) occuring within 5 days | Day 1 Brain CT, Day 5 Brain MRI
  Incidence rate symptomatic intracranial hemorrhage (sICH) occuring within 5 days
Neurologic outcomes evaluated by NIHSS | NIHSS should be scored every visit
  Neurologic outcomes evaluated by NIHSS
Neurologic outcomes evaluated by Barthel Index | Day 0, Day 5, Week 12, Early Termination
  Neurologic outcomes evaluated by Barthel Index
The rate of death due to any cause | it is expected that a follow-up for up to 30 days after the last visit.
  The rate of death due to any cause
Incidence rate of adverse events and adverse drug reactions | it is expected that a follow-up for up to 30 days after the last visit.
  Incidence rate of adverse events and adverse drug reactions
Incidence rate of major systemic bleeding according to the International Society on Thrombosis and Hemostasis (ISTH | Laboratory tests (hematological test, clinical chemistry test, urinalysis etc.)- Day 1, Day 3, Day-5, Week 4, Week 12
  Incidence rate of major systemic bleeding according to the International Society on Thrombosis and Hemostasis (ISTH

CONTACTS AND LOCATIONS:
Overall Officials: Jong Sung Kim, MD, Phd, Principal Investigator — Department of Neurology, Asan Medical Center, Seoul, South Korea
Locations (8):
- South Korea (8):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Myongji Hospital, Gyeonggi-do
  - Inje University Busan Paik Hospital, Pusan
  - Asan Medical Center, University of Ulsan, Seoul
  - Korea University Guro Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Soonchunhyang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JS, Lee KB, Park JH, Sung SM, Oh K, Kim EG, Chang DI, Hwang YH, Lee EJ, Kim WK, Ju C, Kim BS, Ryu JM; SAFE-TPA Investigators. Safety and Efficacy of Otaplimastat in Patients with Acute Ischemic Stroke Requiring tPA (SAFE-TPA): A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study. Ann Neurol. 2020 Feb;87(2):233-245. doi: 10.1002/ana.25644. Epub 2019 Nov 29. PMID 31721277